CLINICAL TRIAL: NCT05349370
Title: Lactate Kinetics in Patients Treated for Septic Shock
Brief Title: Lactate Kinetics in Septic Shock
Acronym: LKISS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Region Stockholm (Other Government); European Society of Intensive Care Medicine (Other); The Scandinavian Society of Anaesthesiology and Intensive Care Medicine (SSAI) (Unknown)
Responsible Party: Principal Investigator, Jonathan Grip, Principal Investigator, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K 2022-4066
Record Dates: First submitted 2022-04-22; First posted 2022-04-27 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental): All patients receive the same intervention/sampling protocol
  Interventions: Other: Isotopically labeled lactate

INTERVENTIONS:
Other: Isotopically labeled lactate — A bolus dose of isotopically labeled lactate is given and blood samples from existing catheters are drawn

SUMMARY:
Lactate kinetics will be studied in hospitalized septic patients using a bolus injection of stable isotopically labeled lactate.

DETAILED DESCRIPTION:
Adult septic patients admitted to the Intensive Care Unit (ICU) or Intermediary Medical Unit in Karolinska University Hospital will be recruited within 72 hours from start of symptoms.

Other than fulfilling the definition for sepsis-3, patients need to be equipped with an arterial catheter to be eligible for inclusion. After informed consent (from next of kin when applicable) baseline blood samples are drawn from existing catheter and the subject is given a bolus dose of 20umol/kg 13C-labeled lactate in 20 ml isotonic saline. After this a total of 14 blood samples á 2 ml is drawn in the following 120 minutes. All blood samples are centrifuged and stored in -800 C until analysis. After all subjects have been included sampled are thawed and analyzed for content of endogenous and labeled lactate. Through analysis between their relationship the lactate production and consumption can be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis
* Age >17 years
* Arterial catheter
* Lactate > 2 mmol at any time point prior to inclusion

Exclusion Criteria:

* Mitochondrial defect
* Degenerative muscle disease
* Terminal liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole body rate of appearance of lactate | 2 hours
  The total amount of lactate produced per unit of time

SECONDARY OUTCOMES:
Clearance of lactate | 2 hours
  Amount of plasma that is cleared from lactate per unit of time

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grip J, Falkenstrom T, Promsin P, Wernerman J, Norberg A, Rooyackers O. Lactate kinetics in ICU patients using a bolus of 13C-labeled lactate. Crit Care. 2020 Feb 10;24(1):46. doi: 10.1186/s13054-020-2753-6. PMID 32041652